CLINICAL TRIAL: NCT00210418
Title: Prevention or Cure: A Comparison of the Effectiveness of Targeting Food Supplements to Malnourished Children Compared to Universal Targeting of Children Under Two in Haiti
Brief Title: Effectiveness of Targeting Food Aid to Malnourished Children Compared to Targeting All Children Under Two Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Cornell University (Other); Food and Nutrition Technical Assistance Project (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); World Vision (Other); Government of Germany (Other Government); United Nations World Food Programme (WFP) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 212620-0S-IFPRI; 81051898
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Malnutrition
Keywords: Malnutrition; Infant nutrition; Food, fortified; Growth; Randomized controlled trials; Evaluation studies; Haiti
MeSH Terms: conditions — Malnutrition | interventions — Educational Status

ARMS (2):
- Preventive targeting (Experimental): This arm targeted pregnant and lactating women as well as children 6-23.9 months of age to receive BCC and food assistance. A total of 27 months of enrollment in this program arm was possible.
  Interventions: Dietary Supplement: Fortified food rations; Behavioral: Education and communication to improve feeding practices
- Recuperative targeting (Active Comparator): This arm targeted pregnant and lactating women as well as mothers of malnourished children (WAZ <-2 zscores) between 6 and 59 months of age. A total of 18 months of enrollment was possible in this program arm.
  Interventions: Dietary Supplement: Fortified food rations; Behavioral: Education and communication to improve feeding practices

INTERVENTIONS:
Dietary Supplement: Fortified food rations — The Fortified food rations were included in both arms, but targeted to all children 6-24 months of age in the 'preventive' arm and to malnourished children (WAZ <-2 Z-scores) in the 'recuperative arm. Food rations included Corn-Soy Blend, lentils, oil and wheat.
Behavioral: Education and communication to improve feeding practices — The education and communication to improve infant and young child feeding was an integral part of the intervention. In the preventive arm, this intervention was targeted to pregnant and lactating mothers and mothers of children 0-24 months of age. The education was done using mother's groups In the recuperative arm, the BCC intervention was only targeted to pregnant and lactating women and mothers of malnourished children under the age of five.

SUMMARY:
The objective of this study is to compare two approaches to targeting donated supplementary food to young children. The study compares the effectiveness of the widely-used curative approach where targeting is based on the child's poor nutritional status to a preventive approach which targets children in poor communities solely on the basis of age and provides supplementary food to all children aged 6-23 months. Cost-effectiveness of the two targeting approaches will also be assessed.

DETAILED DESCRIPTION:
Under-nutrition is widespread among young children in poor countries. In many countries one of the programmatic responses has been distribution of supplementary food to under-nourished children and, often, their families. Traditionally, children under five years have been identified based on low weight-for-age or other anthropometric indicators, and those below a certain cut-off have received supplements. Typically this results in supplementation of many children in the 3-5 year age range, since they are most likely to display cumulative deficits in height and weight, and thus fall below the chosen cut-off.

However, there has been increasing evidence that the most effective period to ensure benefit from supplementary food is when children are 6 to 24 months of age. This is the period of highest growth velocity among humans and thus a period when most growth faltering occurs.

Based on this evidence, the current study aims to assess the effectiveness and cost-effectiveness of a preventive approach that targets children under 24 months as compared to the traditional "curative" approach that targets malnourished (and usually older) children under the age of 5 years.

The comparison is made in the programmatic context of a US Title II food aid distribution program implemented by an international non-governmental organization in rural Haiti. This programmatic context is common in many countries that receive assistance from the United States Agency for International Development and other donors. The study has also involved development of new nutrition education materials and tools, aimed at enabling caregivers to prevent malnutrition. In addition, a range of program operational issues will be studied in order to yield results useful to other implementers of similar interventions.

Comparison: Comparisons will be made at the level of the program site, with service delivery points randomized either to target food supplements as in the past, based on the child's nutritional status, or to target preventively based on age. Pregnant women and lactating women with infants under 6 months of age will receive supplements under both targeting models. Effectiveness will be assessed based on two cross-sectional surveys, at baseline and two years after full implementation of the program.

ELIGIBILITY:
Inclusion Criteria:

* Family resides in community served by World-Vision Haiti's Maternal and Child Health and Nutrition Program

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2002-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Mean z-scores (height-for-age, weight-for-age, weight-for-height) two years after intervention implemented
Prevalence of undernutrition (stunting, wasting, underweight) two years after implementation of intervention

SECONDARY OUTCOMES:
Maternal knowledge about child feeding practices recommended through behavioral intervention at 2 years after implementation of intervention;
Feeding practices and other caregiving practices at 2 years after implementation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marie T. Ruel, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- World Vision-Haiti, Hinche, Haiti

REFERENCES:
- [Result] Ruel MT, Menon P, Loechl C, Pelto G. Donated fortified cereal blends improve the nutrient density of traditional complementary foods in Haiti, but iron and zinc gaps remain for infants. Food Nutr Bull. 2004 Dec;25(4):361-76. doi: 10.1177/156482650402500406. PMID 15646314
- [Result] Ruel MT, Menon P, Habicht JP, Loechl C, Bergeron G, Pelto G, Arimond M, Maluccio J, Michaud L, Hankebo B. Age-based preventive targeting of food assistance and behaviour change and communication for reduction of childhood undernutrition in Haiti: a cluster randomised trial. Lancet. 2008 Feb 16;371(9612):588-95. doi: 10.1016/S0140-6736(08)60271-8. PMID 18280329
- [Result] Menon P, Ruel MT, Loechl C, Pelto G. From research to program design: use of formative research in Haiti to develop a behavior change communication program to prevent malnutrition. Food Nutr Bull. 2005 Jun;26(2):241-2. doi: 10.1177/156482650502600210. No abstract available. PMID 16060227
- [Result] Menon P, Mbuya M, Habicht JP, Pelto G, Loechl CU, Ruel MT. Assessing supervisory and motivational factors in the context of a program evaluation in rural Haiti. J Nutr. 2008 Mar;138(3):634-7. doi: 10.1093/jn/138.3.634. PMID 18287379
- [Result] Donegan S, Maluccio JA, Myers CK, Menon P, Ruel MT, Habicht JP. Two food-assisted maternal and child health nutrition programs helped mitigate the impact of economic hardship on child stunting in Haiti. J Nutr. 2010 Jun;140(6):1139-45. doi: 10.3945/jn.109.114272. Epub 2010 Apr 14. PMID 20392883